CLINICAL TRIAL: NCT06385327
Title: A Phase 1a/1b, Blinded, Placebo-Controlled Study of the Safety, Tolerability and Pharmacokinetics of Single- and Multiple-Ascending Doses of ABI-5366 in Healthy Subjects and in Subjects Who Are Seropositive for Herpes Simplex Virus Type 2 With Recurrent Genital Herpes
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Antiviral Activity of ABI-5366 in Healthy Participants and Participants Seropositive for HSV-2 With Recurrent Genital Herpes
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABI-5366-101
Record Dates: First submitted 2024-04-18; First posted 2024-04-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Genital Herpes Simplex Type 2
Keywords: ABI-5366; PK; Healthy Participants; HSV-2; Recurrent Genital Herpes
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part A: SAD Cohorts 1-5, ABI-5366 (Experimental): Single dose of ABI-5366 (tablet) in Part A for Cohorts 1-5
  Interventions: Drug: ABI-5366; Drug: ABI-5366 Placebo
- Part A: SAD Cohorts 1-5, Placebo (Placebo Comparator): Single dose of matching placebo (tablet) in Part A for Cohorts 1-5
  Interventions: Drug: ABI-5366; Drug: ABI-5366 Placebo
- Part A: SAD Fed Cohort 6, ABI-5366 (Experimental): Single dose of ABI-5366 (tablet) in Part A for Cohort 6, food effect
  Interventions: Drug: ABI-5366
- Part B: MAD Cohorts 1-4 ABI-5366 (Experimental): Weekly or monthly dose of ABI-5366 (tablet) in Part B for Cohorts 1-4. May have a loading dose.
  Interventions: Drug: ABI-5366; Drug: ABI-5366 Placebo
- Part B: MAD Cohorts 1-4 Placebo (Placebo Comparator): Weekly or monthly dose of matching placebo (tablet) in Part B for Cohorts 1-4. May have a loading dose.
  Interventions: Drug: ABI-5366; Drug: ABI-5366 Placebo

INTERVENTIONS:
Drug: ABI-5366 — Once daily tablet dosing (SAD) or weekly or monthly tablet dosing over the 29-day treatment period (MAD)
Drug: ABI-5366 Placebo — Once daily tablet dosing (SAD) or weekly or monthly tablet dosing over the 29-day treatment period (MAD)
  Arms: Part A: SAD Cohorts 1-5, ABI-5366; Part A: SAD Cohorts 1-5, Placebo; Part B: MAD Cohorts 1-4 ABI-5366; Part B: MAD Cohorts 1-4 Placebo

SUMMARY:
This study is designed to assess safety, tolerability, and pharmacokinetics (PK) of single ascending dose (SAD) of ABI-5366 in Part A in healthy participants and multiple-ascending doses (MAD) of ABI-5366 in Part B in participants seropositive for Herpes Simplex Virus Type 2 (HSV-2) with recurrent genital herpes. Effect of food will also be evaluated in Part A.

ELIGIBILITY:
Part A: Inclusion Criteria:

* Subject has a body mass index (BMI) between ≥ 18.0 and < 32.0 kg/m2
* In good health (as determined by the Investigator) based on medical history, physical examination, ECG, and clinical laboratory results.
* Female subjects must be non-pregnant and have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day -1 or Day 1 (predose)
* Agreement to comply with protocol-specified contraceptive requirements

Part B: Inclusion Criteria:

* Subject has a body mass index (BMI) between ≥ 18.0 and < 32.0 kg/m2
* Other than HSV infection, is in good health (as determined by the Investigator) based on medical history, physical examination, ECG, and clinical laboratory results.
* Female subjects must be non-pregnant and have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day 1 (predose)
* Agreement to comply with protocol-specified contraceptive requirements

Part A and B: Exclusion Criteria:

* Current infection of human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), acute hepatitis A virus (HAV), or acute hepatitis E virus (HEV).
* History of any illness that, in the opinion of the Investigator, might confound the results of the study, pose an additional risk in administering study drug to the subject, or a condition known to interfere with the absorption/distribution/elimination of drugs.
* History of any significant drug-related allergic reactions such as anaphylaxis, Stevens-Johnson syndrome, urticaria, or multiple drug allergies
* History of persistent alcohol abuse or illicit drug abuse within 3 years prior to Screening
* Has participated in a clinical study involving administration of either an investigational or a marketed drug within 30 days or 5 half-lives before Screening, whichever is longer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Time Curve (AUC) of ABI-5366 | SAD Cohorts: before and at pre-specified time points up to 168 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Maximum Observed Plasma Concentration (Cmax) of ABI-5366 | SAD Cohorts: before and at pre-specified time points up to 168 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Time to Cmax (Tmax) of ABI-5366 | SAD Cohorts: before and at pre-specified time points up to 168 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Apparent Terminal Elimination Half Life (t 1/2) of ABI-5366 | SAD Cohorts: before and at pre-specified time points up to 168 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Apparent Systemic Clearance (CL/F) of ABI-5366 | SAD Cohorts: before and at pre-specified time points up to 168 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Apparent Volume of Distribution (Vz/F) of ABI-5366 | SAD Cohorts: before and at pre-specified time points up to 168 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Dose normalized AUCs and Cmax of ABI-5366 | SAD Cohorts: before and at pre-specified time points up to 168 hours after dosing. MAD Cohorts: before and at pre-specified time points up to 8 hours after dosing.
Proportion of subjects with adverse events (AEs), premature treatment discontinuation due to AEs, and abnormal laboratory results | Up to 98 days after last dose

SECONDARY OUTCOMES:
SAD Cohorts: Comparison of plasma AUC and Cmax between fasted and fed treatments | SAD Cohorts: before and at pre-specified time points up to 168 hours after dosing.
MAD Cohorts: If applicable, comparison of plasma PK profiles and parameters with and without loading doses | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in viral shedding rate (number of anogenital swabs positive for HSV-2 DNA/total number of swabs) across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in mean and median HSV-2 DNA copies/mL for swab samples positive for HSV-2 DNA across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in the proportion of swab samples with HSV-2 DNA >4 log10 copies/mL across treatments (number of swabbing samples with HSV-2 DNA >4 log10 copies/mL / total number of swabs obtained) | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in number of shedding episodes during the swabbing period across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in duration of shedding episodes during the swabbing period across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in subclinical shedding rate (number of swabs positive for HSV-2 DNA in the absence of lesions/total number of swabs in the absence of lesions) across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in lesion rate during the swabbing period across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in lesion duration during the swabbing period across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.
MAD Cohorts: Difference in recurrence rate (number of reappearances of lesions during the swabbing period/total days assessed) across treatments | MAD Cohorts: At pre-specified time points from Days 8 to 36.

CONTACTS AND LOCATIONS:
Locations (15):
- Australia (7):
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Canopy Clinical Sutherland, Miranda, New South Wales
  - Momentum Clinical Research, Sydney, New South Wales
  - Canopy Beaches Clinical Research, Sydney, New South Wales
  - Canopy Clinical Wollongong, Wollongong, New South Wales
  - Momentum Sunshine, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- New Zealand (8):
  - New Zealand Clinical Research, Auckland
  - New Zealand Clinical Research Christchurch, Christchurch
  - Pacific Clinical Research Network - Hamilton, Hamilton
  - Pacific Clinical Research Network - Tasman, Nelson
  - Momentum Palmerston North, Palmerston North
  - Pacific Clinical Research Network - Rotorua, Rotorua
  - Pacific Clinical Research Network - Wellington, Upper Hutt
  - Momentum Kapiti, Waikanae

IPD SHARING:
Plan to Share IPD: No